CLINICAL TRIAL: NCT05854030
Title: A Study on Serum Exosomal miRNA Predicting the Effective and Prognosis of Immunotherapy Combined With Chemotherapy in Pulmonary Squamous Carcinoma
Brief Title: Serum Exosomal miRNA Predicting the Therapeutic Efficiency in Lung Squamous Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Tianjin Chest Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCC-EV-2022
Record Dates: First submitted 2023-04-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-03

CONDITIONS: Lung Neoplasm; Squamous Cell Carcinoma; Exosomes
Keywords: biomarker
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- advanced lung squamous carcinoma: advanced pulmonary carcinoma with pathological diagnosis of squamous cell and are applied with first line treatment of anti-PD-L1 combined with chemotherapy
  Interventions: Diagnostic Test: collect plasma samples and clinical features
- normol volunteers: 10 normol volunteers will be enrolled in the group
  Interventions: Diagnostic Test: collect plasma samples and clinical features

INTERVENTIONS:
Diagnostic Test: collect plasma samples and clinical features — 8ml of peripheral blood need to be collected from pre- and post-treatment advanced pulmonary squamous carcinoma separately

SUMMARY:
This is an observational prospective bi-center study of 50 patients operated on advanced squamous cell carcinoma. The main aim is to investigate the efficacy of serum exosomal miRNA as a biomarker for predicting the therapeutic effect of immunotherapy combined with chemotherapy.

DETAILED DESCRIPTION:
PD-L1 Testing in guiding patient selection for PD-1/PD-L1 inhibitor therapy in Lung Cancer exhibits insufficient sensitivity and efficacy. The investigators aimed to identify specific serum exosomal miRNA biomarkers that are highly sensitive and stable for predicting the therapeutic effect of immunotherapy combined with chemotherapy. So that the clinicians could use the biomarker to better stratify patients and select potential immunotherapy-beneficial subgroups before clinical decisions.

We plan to enroll 50 patients with advanced treatment-naïve squamous cell carcinoma and 10 healthy people in the present study. Peripheral blood from the plasma of 10 healthy individuals and 50 pulmonary squamous cell carcinoma (SCC) patients will be collected before first-line treatment and after 2 cycles of anti-PD-L1 immunotherapy combined with chemotherapy.

Firstly, exosomal miRNAs extracted from peripheral blood will be analyzed through high-throughput RNA sequencing to identify specific exosomal miRNAs.

Secondly, through analyzing the PFS and OS follow-up data of patients, they are divided into different subgroups. We explore the value of early predicting efficacy of exosome miRNA basing on sequencing results.

Thirdly, we compared the exo-miRNA biomarker with the value of PD-L1 expression in predicting the efficacy of immunotherapy.

Lastly, we suggest exo-miRNA combined with PD-L1 as a biomarker combination in predicting anti-PD-L1 immunotherapy efficacy to better select the potential benefit population suitable for immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histology or cytology confirmed patients with stage IV squamous cell carcinoma of IASLC TNM (8th edition);
2. Patients have not previously received first-line anti-tumor systemic therapy for advanced lung cancer;
3. At least one measurable lesion according to the irRECIST 1.1 standard;
4. Physical condition and organ function allow for systemic antitumor therapy, including standard chemotherapy and immunotherapy;
5. Age ≥ 18 years at the time of signing the informed consent form;
6. Estimated survival≥ 3 months;
7. Patients can follow the planned schedule and actively cooperate in returning to the hospital for regular clinical follow-up and necessary treatment;
8. It can provide the clinical data required for research and is willing to use the test data for further scientific research and commercial product development.

Exclusion Criteria:

1. Other malignancies within the last 5 years (except adequately treated carcinoma in situ and basal or squamous cell skin cancer);
2. The investigators judged that the patient also had other serious medical conditions that could affect follow-up and short-term survival;
3. Any other medical condition and social/psychological problems which the investigator determines that the patient is not suitable to participate in this study;
4. Contrast-enhanced MRI or contrast-enhanced CT for clinical follow-up is not acceptable;
5. Have an active or previous auto-immune disease that is likely to recur;
6. Other antineoplastic therapies were planned for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as advanced lung squamous carcinoma by histopathology and be treated with anti-PD-L1 combined with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
plasma exosomal miRNA level | Baseline up to 21 days
  The expression levels of serum exosome micro RNA
PD-L1 | Baseline up to 21 days
  the expression levels of PD-L1
Imaging data of lesions | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Imaging data of the pulmonary and metastatic lesions of the patients are collected
Objective response rate | From the start of systemic treatment date until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Richeng Richeng, Postdoctor, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walsh RJ, Soo RA. Resistance to immune checkpoint inhibitors in non-small cell lung cancer: biomarkers and therapeutic strategies. Ther Adv Med Oncol. 2020 Jul 3;12:1758835920937902. doi: 10.1177/1758835920937902. eCollection 2020. PMID 32670423
- [Result] Hansen AR, Siu LL. PD-L1 Testing in Cancer: Challenges in Companion Diagnostic Development. JAMA Oncol. 2016 Jan;2(1):15-6. doi: 10.1001/jamaoncol.2015.4685. No abstract available. PMID 26562503
- [Result] Sacher AG, Gandhi L. Biomarkers for the Clinical Use of PD-1/PD-L1 Inhibitors in Non-Small-Cell Lung Cancer: A Review. JAMA Oncol. 2016 Sep 1;2(9):1217-22. doi: 10.1001/jamaoncol.2016.0639. PMID 27310809
- [Result] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Result] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Result] Yu W, Hurley J, Roberts D, Chakrabortty SK, Enderle D, Noerholm M, Breakefield XO, Skog JK. Exosome-based liquid biopsies in cancer: opportunities and challenges. Ann Oncol. 2021 Apr;32(4):466-477. doi: 10.1016/j.annonc.2021.01.074. Epub 2021 Feb 4. PMID 33548389
- [Result] Mashouri L, Yousefi H, Aref AR, Ahadi AM, Molaei F, Alahari SK. Exosomes: composition, biogenesis, and mechanisms in cancer metastasis and drug resistance. Mol Cancer. 2019 Apr 2;18(1):75. doi: 10.1186/s12943-019-0991-5. PMID 30940145
- [Result] Correction: Correlation of plasma exosomal microRNAs with the efficacy of immunotherapy in EGFR / ALK wild-type advanced non-small cell lung cancer. J Immunother Cancer. 2020 May;8(1):e000376corr1. doi: 10.1136/jitc-2019-000376corr1. No abstract available. PMID 32434787
- [Result] Cazzoli R, Buttitta F, Di Nicola M, Malatesta S, Marchetti A, Rom WN, Pass HI. microRNAs derived from circulating exosomes as noninvasive biomarkers for screening and diagnosing lung cancer. J Thorac Oncol. 2013 Sep;8(9):1156-62. doi: 10.1097/JTO.0b013e318299ac32. PMID 23945385
- [Result] Zhang C, Chong X, Jiang F, Gao J, Chen Y, Jia K, Fan M, Liu X, An J, Li J, Zhang X, Shen L. Plasma extracellular vesicle derived protein profile predicting and monitoring immunotherapeutic outcomes of gastric cancer. J Extracell Vesicles. 2022 Apr;11(4):e12209. doi: 10.1002/jev2.12209. PMID 35362262
- [Result] Cordonnier M, Nardin C, Chanteloup G, Derangere V, Algros MP, Arnould L, Garrido C, Aubin F, Gobbo J. Tracking the evolution of circulating exosomal-PD-L1 to monitor melanoma patients. J Extracell Vesicles. 2020 Jan 7;9(1):1710899. doi: 10.1080/20013078.2019.1710899. eCollection 2020. PMID 32002173